Effect of topical melatonin application on dental implant osseointegration and marginal bone level (Clinical and Radiographic Evaluation)

October 21, 2019

Republic of Iraq Ministry of Higher Education And Scientific Research University of Baghdad College of Dentistry



### **Title**

Effect of topical melatonin application on dental implant osseointegration and marginal bone level (Clinical and Radiographic Evaluation)

# **Proposal thesis**

Submitted to the Department of Periodontics, College of Dentistry/University of Baghdad in Partial Fulfillment of the Requirements for Master's Degree in Periodontics.

By Zaid Mohannad Yasser B.D.S.

Supervised by: Prof. Dr. Saif S.Saliem B.D.S., M.Sc. (Periodontics)

2019-2020

#### Introduction:-

Melatonin (N-acetyl-5-methoxy-tryptamine) is an indoleamine synthesized and secreted by the pineal gland and other organs, such as the retina, bone marrow, and intestines in a circadian pattern. Extrapineal sites contribute poorly, or only upon specific stimuli to circulating melatonin (Hardeland et al., 2006). Melatonin influences numerous physiological actions that may be mediated by the binding of the indoleamine to membrane receptors in all tissues (Girgert et al., 2009). Because of its lipophilic properties, melatonin passes through cell membranes to gain access to subcellular organelles (Hevia et al., 2008), being capable to bind to some cytosolic proteins like kinase-C (Macías et al., 2003). Currently, melatonin is not considered a hormone in the classical sense of the term, because it is synthesized in several organs and does not exert effects on a specific target (Tan et al., 2003), but it is rather a powerful cell protector against molecular damage. For the synthesis of melatonin, the pineal cells take up tryptophan from the blood and, through hydroxylation and a decarboxylation process, turn it into serotonin. Serotonin is then converted into N-acetylserotonin through N-acetyltransferase and subsequently methylated to the final form of melatonin by the enzyme hydroxy indole-0-methyltransferase (Reiter, 1991) (Figure 1). In healthy individuals, the maximum secretion of melatonin occurs between midnight and 2 a.m., then it decreases to a minimum during the day(Simonneaux and Ribelayga, **2003)**. Melatonin has numerous physiological functions in different parts of the body, such as the control of circadian rhythms (McArthur et al., 1997), regulation of body temperature(Dollins et al., 1994), and activation of the immune system(Guerrero and Reiter, 2002). In the oral cavity, melatonin has been recognized as an important substance with paracrine effects on nearby cells(Tresguerres et al., 2002), it also acts as an antioxidant and an antiinflammatory and plays an important role in bone formation and in the reduction of bone resorption(Peyrot et al., 2008, Hardeland et al., 2009).



Figure 1. Melatonin synthesis and representation of its molecule (Reiter, 1991)

Osseointegration defined as a direct connection between living bone tissues and a titanium implant without any connective tissues. Osteoblasts are bone formative cells, and osteoclasts are bone resorptive cells. When these cells work together physiologically, the formation and resorption processes of bone tissue is known as bone remodelling. The remodeling of bone tissues is regulated by the action of systemic hormones (estradiol, parathyroid, growth, and melatonin) and by the bone marrow and osteoid matrix-derived growth factors(Tresguerres et al., 2012, Wulandari). Insufficient bone quality and quantity can be seen frequently in elderly populations with atrophic and osteoporotic bones, and this situation stems from increased osteoclastic activity due to a reduction in osteoblastogenesis. In addition, local free radical concentrations in all body cells, including osteoblasts, can reduce osteoblastic activity in aged patients. This process could lead to a reduction in bone regeneration capacity(Cao et al., 2005). Melatonin can also suppress osteoclastogenesis, and therefore inhibit bone tissue

resorption(Cutando et al., 2008, Witt-Enderby et al., 2006). In addition to this, *in vitro* research has reported that melatonin can increase osteoblast proliferation and differentiation (López-Martínez et al., 2012, Muñoz et al., 2012). So was proposed that the local application of melatonin during surgical implant placement procedures would be an effective treatment technique for dental implant osseointegration (Dundar et al., 2016). Worthy osseointegration is a prerequisite for dental implants. Optimal osseointegration depends on the formation of new bone around implants, which may be stimulated by the application of biomimetic agents (Ramazanoglu et al., 2011). Considering the bone metabolism, melatonin acts directly on the osteoclast, a multinucleated cell, which resorbs the extracellular matrix through various mechanisms, including the production of free radicals (Roth et al., 1999). Moreover, in pre-osteoblast cultures from rats, melatonin, in a dose-dependent manner, promoted the development of bone sialoprotein and other protein bone markers, including alkaline phosphatase, osteopontin, and osteocalcin, and speeds up their period of differentiation into osteoblasts from the normal rate, which is 21 days, to 12 days, this reaction is mediated by the membrane receptors for the indole (Roth et al., 1999). Also, melatonin, may interfere with the function of the osteoclast and thereby inhibit bone resorption(Cardinali et al., 2003). (Cutando et al., 2008) conducted an experimental study using melatonin with dental implants in dogs. Two weeks after implant insertion, melatonin significantly increased all parameters of osteointegration. It has been observed that melatonin, increases bone mass by suppressing resorption through down-regulation of the RANKLmediated osteoclast formation and activation (Cutando et al., 2007). These data point towards an osteogenic effect of melatonin that may be of clinical importance, as it could be used as a therapeutic agent in situations in which bone formation would be advantageous, such as in the treatment of fractures or of osteoporosis (Cardinali et al., 2003).

### **Toxicology of Melatonin:-**

The physiological functions of the pineal hormone melatonin are extremely diverse. The functions include direct and indirect modulations of anti-oxidative defense, blood pressure, body temperature, cortisol rhythm, reproduction and immune function (Claustrat and Leston, 2015). Correspondingly, exogenous melatonin has been investigated as a treatment for a number of medical and surgical diseases, demonstrating encouraging results (Andersen et al., 2014, Gitto et al., 2011). In the USA, melatonin is available as an over-the-counter nonprescription drug. In most European countries, however, melatonin remains a prescription drug (Circadin) and has only been approved as a treatment for primary insomnia in people over 55 years of age. However, a recent Norwegian register study documented a 3- to 5-times increase in off-label use among children and adolescents in the time period 2004 to 2012 (Hartz et al., 2015). Melatonin is generally considered safe (Yousaf et al., 2010), but the increasing clinical use with potentially increasing doses necessitates further investigations of the risks of both mild and serious adverse effects. In experimental animal studies, exogenously administered melatonin has been given in doses up to 800 mg/kg without any acute toxic effects (Barchas et al., 1967). A number of studies in preterm infants have investigated the anti-oxidative/anti-inflammatory and clinical effects of exogenous melatonin in different conditions, such as pain during tracheal intubation (10 mg/kg x 10 doses, randomized) (Gitto et al., 2012), asphyxia (10 mg x 8 doses, randomized) (Fulia et al., 2001), respiratory distress (10 mg/kg x 10 doses, randomized) (Gitto et al., 2004b). Despite repeated high doses of intravenous melatonin, no signs of adverse effects were observed (Gitto et al., 2004c, Gitto et al., 2004a). Oral melatonin in doses of 0.5-10 mg was administered daily from 10 days to 12 weeks to improve sleep quality (Wright et al., 2011, Cortesi et al., 2012). The studies performed detailed registration of possible adverse effects, demonstrating a number of mild adverse effects, such as agitation, dizziness, headache, nausea, and sleepiness (Wasdell et al., 2008, Jain et al., 2015). Another study was to assess the toxicology of melatonin (10 mg), administered for 28 days to 40 volunteers randomly assigned to groups receiving either melatonin (N\_30) or placebo (N\_10) in a double-blind fashion, according to

the parameters analyzed, there is no toxicological effect that might compromise the use of melatonin at a dose of 10 mg for the period of time utilized in this study(Seabra et al., 2000). A randomized, double-blind, placebo-controlled study including 54 female patients undergoing breast cancer surgery were given 6 mg of oral melatonin or placebo to improve depressive symptoms and anxiety during a three month investigational period (Hansen et al., 2014). Finally, a randomized, double-blind, placebo-controlled study was conducted in elderly patients suffering from Alzheimer's disease who were administered 2 mg of melatonin or placebo for a 24-week period (Wade et al., 2014). A substantial number of both animal and human studies document that short-term use of melatonin is safe, even in extreme doses. No studies indicate that exogenous melatonin possesses any serious adverse effects. Also, randomized clinical studies indicate that long-term administration only induces mild adverse effects comparable to placebo treatment. (Andersen et al., 2016).

#### Periotest M device:-

Periotest device was developed to measure the damping characteristics of natural teeth and has been used to evaluate implant (Cehreli et al., 2009). It was developed by Schulte in 1983 to quantify TM (Shulte et al., 1983), and then utilized by Teerlinck et al. (1991), to measure implant stability and to overcome destructive methods in measuring the implant stability like histologic analysis, tensional test, push-out/pull-out test and removal torque analysis. The (Classic/Wired) Periotest device has been the subject of several studies with generally favorable results. These results showed that the Periotest device generally demonstrated a high degree of repeatability and reliability. A wireless version of the Periotest (Periotest "M") has been introduced to the profession. According to information provided by the electronic page of the Periotest M /wireless device manufacturer (Medizintechnik Gulden, Modautal, Germany), Periotest M is simpler to perform an objective evaluation of an implant's stability compared to classic Periotest. In Periotest M wireless design, the user can benefit from maximum freedom of movement. The device can be used for taking measurements on a wide variety of implants, without the need for any special accessories, such as a smart peg (Pang et al., 2014). The Periotest has an

important advantage against the others like the Osstell device: it can be applied directly to the implant superstructure (Geckili et al., 2009).

The limitations of Periotest are the inability of the instrument to measure the mesiodistal mobility, the possible effect of position and angle of the rods on the measured value (Satwalekar et al., 2015). The readings of PTV are from (–8 to +50) according to information provided by the device manufacturer (Medizintechnik Gulden, Modautal, Germany) (Pang et al., 2014), (Table 1). These readings are displayed digitally on a monitor as (PTVs), (Aparicio et al., 2006).

(Table 1): Interpretation of readings of implant stability in periotest (Pang et al., 2014).

| Reading | Interpretation |
|---|---|
| -8 to 0.0 | Good osseointegration, the implant can be loaded. |
| +0.1 to +9.9 | Clinical examination is required, in most cases, loading is not possible. |
| +10 to +50 | Osseointegration is not sufficient, the implant cannot be loaded. |

# Cone-beam computed tomography (CBCT):-

Cone-beam computed tomography (CBCT) is an imaging modality that offers significant advantages for the evaluation of implant patients (Hatcher et al., 2003, Schulze et al., 2005). The field of view (FOV) is an important feature that describes the extent of the imaged volume from large FOV (greater than 15 cm) to medium FOV (8 to 15 cm) and limited FOV (less than 8 cm). Limited FOV units image a small area, delivering less radiation and producing a higher-resolution image (Newman et al., 2018). CBCT allows for defining with elevated accuracy the quality (cortical/medullar ratio) and the quantity (height and thickness) of bone available for the implant, providing the essential information of performing or not a preimplant bony graft (Garlaschi et al., 2014). when compared to medical CT, CBCT can be recommended as a dose reducing technique for dental

implant applications (**Okano et al., 2009, Qu et al., 2010**). The effective dose from CBCT examinations ranges from 13  $\mu$  Sv with the 3D Accuitomo CBCT machine using the 4 x4 cm FOV to 479  $\mu$  Sv with the CB Mercury CBCT machine (**Table 2**). For comparison, the effective dose from one panoramic radiograph is approximately 10 to 14 $\mu$ Sv(**Ludlow et al., 2006**). Furthermore, the exposure from a maxillomandibular medical CT ranges from 474 to 1160  $\mu$ Sv(**Loubele et al., 2009**). The average background radiation in the United States is 3000  $\mu$ Sv (3 mSv) per year or 8  $\mu$ Sv per day (**Table 2**). It is important to understand that every effort must be made to reduce the effective radiation dose to the patient. By using the smallest possible FOV, the lowest mA setting, the shortest exposure time, and a pulsed exposure mode of acquisition, it is possible to accomplish effective dose reduction to the patient(**Sur et al., 2010**).

| CBCT<br>Scanner | FOV (cm) | Effective Dose<br>(µSv) | Digital Panoramic<br>Equivalent (14 μSv) | No. of Days of Annual<br>per Capita Background<br>(3 μSv = 3000 μSv) | References |
|---|---|---|---|---|---|
| | 22/13 (40 s)/13 (10 s) | 82/77/48 | 5.9/5,5/3.4 | 10/9,4/5.8 | Loubele et al10 |
| | 6 min. (low resolution/<br>high resolution) | 96.2/118.5 | 6.9/8.5 | 11.7/14.4 | Hatcher <sup>20</sup> |
| | 6 max, (low resolution/<br>high resolution) | 58.9/93,3 | 4.2/6.6 | 7.2/11 | Hatcher <sup>20</sup> |
| | 22/13 | 206.2/133.9 | 14.7/9.6 | 25/16 | Hatcher <sup>20</sup> |
| | 13 | 61.1 | 4.4 | 7.4 | Silva et al <sup>21</sup> |
| -CAT next<br>generation | 23 × 17 | 74 | 5.3 | 9 | Ludlow and<br>Ivanovic <sup>15</sup> |
| | 16 × 13 (19 mAs) | 87 | 6.2 | 10.6 | Ludlow and<br>Ivanovic <sup>15</sup> |
| | 16 × 13 (18.5 mAs) | 83 | 5.9 | 10.2 | Pauwels at aPI |
| | 16 × 6 | 45 | 3.2 | 5.5 | Pauwels et al? |
| Newtorn 9000 | 23 | 56.2 | 4 | 6.9 | Silva et al21 |
| | 12 in (male/female) | 93/95 | 6.6/6.8 | 11.3/11.6 | Coppenrath<br>et al <sup>20</sup> |
| Newtorn 3G | 19 | 68 | 4.9 | 8.3 | Ludlow and<br>Ivanovic <sup>16</sup><br>Ivanovic <sup>16</sup> |
| | 8 × 8 (72 mAs/96 mAs) | 488/652 | 35/47 | 59/79 | Ludlow and<br>Ivanovic <sup>15</sup> |
| | 8 × 8 (169 mAs/19.9<br>mAs) | 122/28 | 8.7/2 | 15/1.7 | Pauwels et al <sup>22</sup> |
| Picasso-Trio | 12 × 7 (127 mAs/91<br>mAs) | 123/81 | 8.8/5.8 | 15.1/10 | Pauwels et al <sup>22</sup> |
| PaX-Uni3D | 5 × 5 max. | 44 | 3.1 | 5.4 | Pauwels et al22 |
| Kodak 9000<br>3D | Max. ant./min. post. | 19/40 | 1,4/2.9 | 2.3/4.9 | Pauwels et al <sup>23</sup> |
| | 20 × 18 | 92 | | | Pauwels et al <sup>22</sup> |
| | 15 × 9 | 136 | | | Pauwels et al73 |
| | 20 × 18 (small/medium/<br>large adult) | 76/98/166 | 5.4/7.0/11.9 | 9.3/12.1/20.4 | Ludlow et al <sup>74</sup> |
| | 15 × 9 (small/medium/<br>large adult) | 93/163/260 | 6.6/11.6/18.6 | 11.4/20.1/32.0 | Ludlow et al <sup>24</sup> |
| | 28 mAs | 84 | 6 | 10.3 | Pauwels et al <sup>23</sup> |
| SCANORA 3D | 14.5 × 13 | 68 | 4.9 | 8.4 | Pauwels et al <sup>20</sup> |
| | 10 × 7.5 | 46 | 3,3 | 5.7 | Pauwels et al <sup>27</sup> |
| SkyView . | 17 × 17 | 87 | 6.2 | 10.7 | Pauwels et al <sup>22</sup> |
| ILÚMA | 19 × 19 (20 mAs/152<br>mAs) | 98/498 | 7/36,6 | 11.9/60.6 | Ludlow and<br>Ivanovic <sup>16</sup> |
| | 20.5 × 14 (76 mAs) | 368 | 26.3 | 45.3 | Pauwels et al <sup>12</sup> |

### Aim and objectives:-

**Aim: -** To evaluate the osseointegration following the application of melatonin around dental implants.

### **Objectives: -**

- 1- Measuring primary and secondary stability of the dental implant by Periotest M device.
- 2- Measuring marginal bone level around the dental implant in baseline and after 6 months follow up using a cone-beam computed tomography (CBCT).

### **Research Hypothesis:-**

The topical application of melatonin powder in the osteotomy site has an effect on osseointegration around the dental implant and minimize marginal bone loss.

### Null hypothesis:-

The topical application of melatonin powder in the osteotomy site has no effect on osseointegration around the dental implants and in minimizing marginal bone loss.

### Methodology:-

**Study design:** - a split-mouth clinical trial.

### **Setting & Subjects:**

The study will be conducted in a split-mouth design on patients male with missing teeth in the upper or lower jaw (canine to  $1^{\rm st}$  molar area), the subjects will be selected depending on bone density and from those attending to the department of periodontics.

#### Inclusion criteria:

- 1. Patients male have good oral hygiene.
- 2. Patients were periodontally healthy.
- 3. Patients had at least two missing teeth in the upper or lower jaw (canine to 1st molar area) indicated for the dental implant.

#### **Exclusion criteria:**

- 1-Patients with any systemic diseases that influence bone healing such as osteoporosis and diabetes mellitus.
- 2-Fully edentulous.
- 3-Patients who had parafunctional habits.
- 4-Smokers.
- 5-Patients who were not able to follow the treatment protocol.

### Sample Size:

Twenty single-piece endosseous implants use for patients with at least two missing teeth in the upper or lower jaw (canine to 1st molars area).

#### Materials:-

- 1-Melatonin powder (*N-Acetyl-5-methoxytryptamine*) from (Sigma-Aldrich/Germany).
- 2-Periotest M device (Medizintechnik Gulden, Germany).
- 3-Dentium implant surgical kit system and DI fixtures (Dentium Co., Korea).

#### **Procedure:**

Twenty single-piece endosseous implants (Dentium Co, Korea) will use to restore missing teeth in the upper or lower jaw (canine to 1st molars area) from both sides. The study will be split-mouth technique, each patient serves as his own control (served into 2 groups), the study side (topical application of melatonin in the implant side), and the control side (no melatonin in the other implant side of the same patients). According to the study reported by (Cutando et al., 2008) the estimated dose of melatonin required to enhance osseointegration of dental implant and minimize the marginal bone resorption is 1.2 mg of melatonin powder for each implant. CBCT for all patients before implant placement to determine bone density, dimension, and anatomical landmarks. Prior to surgery, all patients will instruct to use chlorhexidine 0.12% mouthwash as antiseptic. After local anesthesia, a mucoperiosteal flap will reflect. The manufacturer's instructions should be followed for the preparation of the implant osteotomy site. For the study

side, 1.2 mg of melatonin powder will place in the osteotomy site before the insertion of the implant. For the control side, no melatonin powder will be used and implants will be inserted directly in the prepared implant site. After dental implant installation, the gingival former will insert into the body of the fixture, then the Periotest M device will use to measure the primary stability of the DI fixture. After that, the gingival former will be removed and cover screw place and tightened into the fixture. Sutures will place after flap replacement. Patients should be instructed to use antibiotics amoxicillin 500mg and metronidazole 500mg 3 times/day for 5 days after surgical procedure, soft diet and proper oral hygiene measures. Also, CBCT immediately after implant placement to record baseline bone level, CBCT after 6 months follow up to measure marginal bone level around implant comparing with baseline measurement, and measure the secondary stability using periotest M device.

### **Stopping rules**

The occurrence of an unexpected include implant failure...

# **Budget and funding**

This study is self-funded.

# Justification for ethical approval:-

According to the college of the dentistry/university of Baghdad following the Declaration of Helsinki / Tokyo on medical protocol and ethics.

#### Dissemination

Postgraduate Thesis.

#### References

ANDERSEN, L., WERNER, M., ROSENBERG, J. & GÖGENUR, I. 2014. A systematic review of peri-operative melatonin. *Anaesthesia*, 69, 1163-1171

ANDERSEN, L. P. H., GÖGENUR, I., ROSENBERG, J. & REITER, R. J. 2016. The safety of *investigation*, 36, 169-175 melatonin in humans. Clinical drug

BARCHAS, J., DACOSTA, F. & SPECTOR, S. 1967. Acute pharmacology of melatonin. CAO, J. J., WRONSKI, T. J., IWANIEC, U., .*Nature*, 214, 919

PHLEGER, L., KURIMOTO, P., BOUDIGNON, B. & HALLORAN, B. P. 2005. Aging increases stromal/osteoblastic cell-induced osteoclastogenesis and alters the osteoclast precursor pool in the mouse. *Journal of Bone and Mineral Research*, 20, 1659-1668

CARDINALI, D. P., LADIZESKY, M. G., BOGGIO, V., CUTRERA, R. A. & MAUTALEN, C. 2003. Melatonin effects on bone: experimental facts and clinical perspectives. *Journal of pineal research*, 34, 81-87

CLAUSTRAT, B. & LESTON, J. 2015. Melatonin: Physiological effects in humans. *Neurochirurgie*, 61, 77-84

VALENTE, D. 2012. & .CORTESI, F., GIANNOTTI, F., SEBASTIANI, T., PANUNZI, S Controlled-release melatonin, singly and combined with cognitive behavioural therapy, for persistent insomnia in children with autism spectrum disorders: a .randomized placebo-controlled trial. *Journal of sleep research*, 21, 700-709

CUTANDO, A., GóMEZ-MORENO, G., ARANA, C., ACUÑA-CASTROVIEJO, D. & REITER, R. J. 2007. Melatonin: potential functions in the oral cavity. *Journal of periodontology*, .78, 1094-1102

CUTANDO, A., GÓMEZ-MORENO, G., ARANA, C., MUñOZ, F., LOPEZ-PEñA, M., J. & REITER, R. J. 2008. Melatonin stimulates osteointegration of 'STEPHENSON dental implants. *Journal of Pineal Research*, 45, 174-179

DOLLINS, A. B., ZHDANOVA, I. V., WURTMAN, R. J., LYNCH, H. J. & DENG, M. H. 1994. Effect of inducing nocturnal serum melatonin concentrations in daytime on sleep, mood, body temperature, and performance. *Proceedings of the National .Academy of Sciences*, 91, 1824-1828

DUNDAR, S., YAMAN, F., SAYBAK, A., OZUPEK, M. F., TOY, V. E., GUL, M. & OZERCAN, İ. H. topical melatonin application on osseointegration 2016. Evaluation of effects of of dental implant: an experimental study. *Journal of Oral Implantology*, 42, 386-.389

EL-GAMMAL, M. Y., SALEM, A. S., ANEES, M. M. & TAWFIK, M. A. 2016. Clinical and radiographic evaluation of immediate loaded dental implants with local application of melatonin: a preliminary randomized controlled clinical trial. *.Journal of Oral Implantology*, 42, 119-125

FULIA, F., GITTO, E., CUZZOCREA, S., REITER, R. J., DUGO, L., GITTO, P., BARBERI, S., CORDARO, S. & BARBERI, I. 2001. Increased levels of malondial dehyde and

- nitrite/nitrate in the blood of asphyxiated newborns: reduction by melatonin. *Journal of pineal research*, 31, 343-349
- GIRGERT, R., HANF, V., EMONS, G. & GRUNDKER, C. 2009. Membrane-bound melatonin receptor MT1 down-regulates estrogen responsive genes in breast cancer cells. *Journal of pineal research*, 47, 23-31
- GITTO, E., AVERSA, S., REITER, R. J., BARBERI, I. & PELLEGRINO, S. 2011. Update on the .use of melatonin in pediatrics. *Journal of pineal research*, 50, 21-28
- GITTO, E., AVERSA, S., SALPIETRO, C. D., BARBERI, I., ARRIGO, T., TRIMARCHI, G., REITER, R. J. & PELLEGRINO, S. 2012. Pain in neonatal intensive care: role of .omelatonin as an analgesic antioxidant. *Journal of pineal research*, 52, 291-29
- GITTO, E., REITER, R. J., AMODIO, A., ROMEO, C., CUZZOCREA, E., SABATINO, G., BUONOCORE, G., CORDARO, V., TRIMARCHI, G. & BARBERI, I. 2004a. Early indicators of chronic lung disease in preterm infants with respiratory distress syndrome and their inhibition by melatonin. *Journal of pineal research*, 36, 250-.255
- GITTO, E., REITER, R. J., CORDARO, S. P., LA ROSA, M., CHIURAZZI, P., TRIMARCHI, G., GITTO, P., CALABRÓ, M. P. & BARBERI, I. 2004b. Oxidative and inflammatory parameters in respiratory distress syndrome of preterm newborns: beneficial .effects of melatonin. *American journal of perinatology*, 21, 209-216
- GITTO, E., ROMEO, C., REITER, R. J., IMPELLIZZERI, P., PESCE, S., BASILE, M., ANTONUCCIO, P., TRIMARCHI, G., GENTILE, C. & BARBERI, I. 2004c. Melatonin reduces oxidative stress in surgical neonates. *Journal of pediatric surgery*, 39, .184-189
- GUERRERO, J. M. & REITER, R. J. 2002. Melatonin-immune system relationships. *Current topics in medicinal chemistry*, 2, 167-179
- MADSEN, M. T., HAGEMAN, I., RASMUSSEN, L. S., ·.HANSEN, M. V., ANDERSEN, L. T BOKMAND, S., ROSENBERG, J. & GÖGENUR, I. 2014. Effect of melatonin on depressive symptoms and anxiety in patients undergoing breast cancer surgery: *cancer research and* a randomized, double-blind, placebo-controlled trial. *Breast* .treatment, 145, 683-695
- HARDELAND, R., PANDI-PERUMAL, S. & CARDINALI, D. P. 2006. Melatonin. *The international journal of biochemistry & cell biology*, 38, 313-316
- HARTZ, I., HANDAL, M., TVERDAL, A. & SKURTVEIT, S. 2015. Paediatric Off-Label Use of Melatonin–A Register Linkage Study between the Norwegian Prescription Database and Patient Register. *Basic & clinical pharmacology & toxicology*, 117, .267-273
- A. 'JAIN, S. V., HORN, P. S., SIMAKAJORNBOON, N., BEEBE, D. W., HOLLAND, K., BYARS W. & GLAUSER, T. A. 2015. Melatonin improves sleep in children with epilepsy: a .randomized, double-blind, crossover study. *Sleep medicine*, 16, 637-644
- LóPEZ-MARTÍNEZ, F., OLIVARES PONCE, P. N., GUERRA RODRÍGUEZ, M. & MARTÍNEZ PEDRAZA, R. 2012. Melatonin: bone metabolism in oral cavity. *International journal of dentistry*, 2012

- LOUBELE, M., BOGAERTS, R., VAN DIJCK, E., PAUWELS, R., VANHEUSDEN, S., SUETENS, P., MARCHAL, G., SANDERINK, G. & JACOBS, R. 2009. Comparison between CBCT and MSCT scanners for dentomaxillofacial effective radiation dose of applications. *European journal of radiology*, 71, 461-468
- LUDLOW, J. B., DAVIES-LUDLOW, L., BROOKS, S. & HOWERTON, W. 2006. Dosimetry of 3 G <sup>r</sup> CBCT devices for oral and maxillofacial radiology: CB Mercuray, NewTom .and i-CAT. *Dentomaxillofacial Radiology*, 35, 219-226
- MCARTHUR, A. J., HUNT, A. E. & GILLETTE, M. U. 1997. Melatonin action and signal transduction in the rat suprachiasmatic circadian clock: activation of protein .kinase C at dusk and dawn. *Endocrinology*, 138, 627-634
- MUñOZ, F., LóPEZ-PEñA, M., MIñO, N., GóMEZ-MORENO, G., GUARDIA, J. & CUTANDO, A. 2012. Topical application of melatonin and growth hormone accelerates bone healing around dental implants in dogs. *Clinical implant dentistry and related* .research, 14, 226-235
- RAMAZANOGLU, M., LUTZ, R., ERGUN, C., VON WILMOWSKY, C., NKENKE, E. & SCHLEGEL, K. A. 2011. The effect of combined delivery of recombinant human bone morphogenetic protein-2 and recombinant human vascular endothelial from biomimetic calcium-phosphate-coated implants on °growth factor 16 .osseointegration. *Clinical oral implants research*, 22, 1433-1439
- REITER, R. J. 1991. Pineal melatonin: cell biology of its synthesis and of its physiological .\^-interactions. *Endocrine reviews*, 12, 151
- ROTH, J. A., KIM, B.-G., LIN, W.-L. & CHO, M.-I. 1999. Melatonin promotes osteoblast differentiation and bone formation. *Journal of Biological Chemistry*, 274, 22041-.22047
- SEABRA, M. D. L. V., BIGNOTTO, M., PINTO JR, L. R. & TUFIK, S. 2000. Randomized, double-blind clinical trial, controlled with placebo, of the toxicology of chronic .melatonin treatment. *Journal of pineal research*, 29, 193-200
- SIMONNEAUX, V. & RIBELAYGA, C. 2003. Generation of the melatonin endocrine the complex regulation of melatonin synthesis message in mammals: a review of by norepinephrine, peptides, and other pineal transmitters. *Pharmacological* .reviews, 55, 325-395
- SUR, J., SEKI, K., KOIZUMI, H., NAKAJIMA, K. & OKANO, T. 2010. Effects of tube current on cone-beam computerized tomography image quality for presurgical implant planning in vitro. *Oral Surgery, Oral Medicine, Oral Pathology, Oral Radiology, and .Endodontology,* 110, e29-e33
- TAN, D. X., MANCHESTER, L. C., HARDELAND, R., LOPEZ-BURILLO, S., MAYO, J. C., SAINZ, REITER, R. J. 2003. Melatonin: a hormone, a tissue factor, an autocoid, a & .R. M .paracoid, and an antioxidant vitamin. *Journal of pineal research*, 34, 75-78
- TRESGUERRES, I. F., CLEMENTE, C., BLANCO, L., KHRAISAT, A., TAMIMI, F. & TRESGUERRES, J. A. 2012. Effects of local melatonin application on implant .osseointegration. *Clinical implant dentistry and related research*, 14, 395-399
- TRESGUERRES, I. F., CLEMENTE, C., DONADO, M., GÓMEZ-PELLICO, L., BLANCO, L., ALOBERA, M. A. & TRESGUERRES, J. A. 2002. Local administration of growth

hormone enhances periimplant bone reaction in an osteoporotic rabbit model: an histologic, histomorphometric and densitometric study. *Clinical oral implants research*, 13, 631-636

M., NIR, T., FRYDMAN- 'WADE, A. G., FARMER, M., HARARI, G., FUND, N., LAUDON MAROM, A. & ZISAPEL, N. 2014. Add-on prolonged-release melatonin for cognitive function and sleep in mild to moderate Alzheimer's disease: a 6-month, 'randomized, placebo-controlled, multicenter trial. *Clinical interventions in aging* 

WASDELL, M. B., JAN, J. E., BOMBEN, M. M., FREEMAN, R. D., RIETVELD, W. J., TAI, J., HAMILTON, D. & WEISS, M. D. 2008. A randomized, placebo-controlled trial of controlled release melatonin treatment of delayed sleep phase syndrome and impaired sleep maintenance in children with neurodevelopmental disabilities. *Journal of pineal research*, 44, 57-64

WITT-ENDERBY, P. A., RADIO, N. M., DOCTOR, J. S. & DAVIS, V. L. 2006. Therapeutic treatments potentially mediated by melatonin receptors: potential clinical uses in the prevention of osteoporosis, cancer and as an adjuvant therapy. *Journal of .pineal research*, 41, 297-305

WRIGHT, B., SIMS, D., SMART, S., ALWAZEER, A., ALDERSON-DAY, B., ALLGAR, V., Melatonin . Y. Y. WHITTON, C., TOMLINSON, H., BENNETT, S. & JARDINE, J versus placebo in children with autism spectrum conditions and severe sleep problems not amenable to behaviour management strategies: a randomised controlled crossover trial. *Journal of autism and developmental disorders*, 41, .175-184

WULANDARI, A. Jumlah Sel Osteoklas yang Mengekspresikan Interleukin 1 Beta (IL-1B) Akibat Induksi Gaya Mekanik Ortodonti Dengan Pemberian Natrium Fluorida .(NaF) Secara Topikal

YOUSAF, F., SEET, E., VENKATRAGHAVAN, L., ABRISHAMI, A. & CHUNG, F. 2010. Efficacy and Safety of Melatonin as an Anxiolytic and Analgesic in the Perioperative PeriodA Qualitative Systematic Review of Randomized Trials. *Anesthesiology:* . *The Journal of the American Society of Anesthesiologists,* 113, 968-976

Peyrot, F. and Ducrocq, C., 2008. Potential role of tryptophan derivatives in stress responses characterized by the generation of reactive oxygen and nitrogen species. Journal of pineal research, 45(3), pp.235-246.

Hardeland, R., Tan, D.X. and Reiter, R.J., 2009. Kynuramines, metabolites of melatonin and other indoles: the resurrection of an almost forgotten class of biogenic amines. Journal of pineal research, 47(2), pp.109-126.

Cehreli, M.C., Karasoy, D., Akca, K. and Eckert, S.E., 2009. Meta-analysis of methods used to assess implant stability. International Journal of Oral & Maxillofacial Implants, 24(6).

SHULTE, W., D'HOEDT, B., LUKAS, D., MUHIBRADT, L., SCHOLZ, F. & BRETSCHI, J. 1983. Periotest-neues messverfahren der function des paradontiums. Zahnarzti Mitt, 73, 1229-40.

PANG, K. M., LEE, J. W. & LEE, J. Y. 2014. Clinical outcomes of magnesium-incorporated oxidised implants: a randomised double-blind clinical trial. Clin Oral Implants Res, 25, 616-21.

GECKILI, O., BILHAN, H. & BILGIN, T. 2009. A 24-week prospective study comparing the stability of titanium dioxide grit-blasted dental implants with and without fluoride treatment. Int J Oral Maxillofac Implants, 24, 684-8.

SATWALEKAR, P., NALLA, S., REDDY, R. & CHOWDARY, S. G. 2015. Clinical evaluation of osseointegration using resonance frequency analysis. J Indian Prosthodont Soc, 15(3), 192-9.

PANG, K. M., LEE, J. W. & LEE, J. Y. 2014. Clinical outcomes of magnesium-incorporated oxidised implants: a randomised double-blind clinical trial. Clin Oral Implants Res, 25, 616-21.

APARICIO, C., LANG, N. P. & RANGERT, B. 2006. Validity and clinical significance of biomechanical testing of implant/bone interface. Clin. Oral Imp Res, 17(2), 2-7. Hatcher, D.C., Dial, C. and Mayorga, C., 2003. Cone beam CT for pre-surgical assessment of implant sites. CDA, 31(11), pp.825-834.

Schulze, D., Heiland, M., Blake, F., Rother, U. and Schmelzle, R., 2005. Evaluation of quality of reformatted images from two cone-beam computed tomographic systems. Journal of Cranio-Maxillofacial Surgery, 33(1), pp.19-23.

Newman, M.G., Takei, H., Klokkevold, P.R. and Carranza, F.A., 2018. Newman and Carranza's Clinical Periodontology E-Book. Elsevier Health Sciences.

Garlaschi, G., 2014. Cone Beam CT and 3D Imaging: A Practical Guide. Springer.

Okano, T., Harata, Y., Sugihara, Y., Sakaino, R., Tsuchida, R., Iwai, K., Seki, K. and Araki, K., 2009. Absorbed and effective doses from cone beam volumetric imaging for implant planning. Dentomaxillofacial Radiology, 38(2), pp.79-85.

Qu, X.M., Li, G., Ludlow, J.B., Zhang, Z.Y. and Ma, X.C., 2010. Effective radiation dose of ProMax 3D cone-beam computerized tomography scanner with different dental protocols. Oral Surgery, Oral Medicine, Oral Pathology, Oral Radiology, and Endodontology, 110(6), pp.770-776.